CLINICAL TRIAL: NCT07094750
Title: Impact of Treatment Intensity on Survival, Quality of Life, and Resource Utilization in Medically Less Fit Adults With Acute Myeloid Leukemia and High-Grade Myeloid Neoplasms: A Randomized Pilot Study
Brief Title: Randomization for the Identification of Best Treatment Intensity for Less Fit Adults With Acute Myeloid Leukemia and Myeloid Neoplasms
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RG1125566; NCI-2025-04530 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-07

CONDITIONS: Acute Leukemia of Ambiguous Lineage; Acute Myeloid Leukemia; Myeloid Neoplasm
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Leukemia, Myeloid, Acute | interventions — Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm I (randomized higher-intensity therapy) (Experimental): Patients receive SOC or investigational higher-intensity therapy on a subsequent treatment trial that is at least as intense as 7+3 regimen at the discretion of the treating physician on study. Treatment continues in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection and bone marrow assessments on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Collection; Other: Electronic Health Record Review; Other: Questionnaire Administration
- Arm II (randomized lower-intensity therapy) (Experimental): Patients receive SOC or investigational lower-intensity therapy on a subsequent treatment trial that is less intense than 5+2 regimen at the discretion of the treating physician on study. Treatment continues in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection and bone marrow assessments on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Collection; Other: Electronic Health Record Review; Other: Questionnaire Administration
- Arm III (patient choice higher-intensity therapy) (Active Comparator): Patients receive SOC or investigational higher-intensity therapy on a subsequent treatment trial that is at least as intense as 7+3 regimen according to physician/patient preference on study. Treatment continues in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection and bone marrow assessments on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Collection; Other: Electronic Health Record Review; Other: Questionnaire Administration
- Arm IV (patient choice lower-intensity therapy) (Active Comparator): Patients receive SOC or investigational lower-intensity therapy on a subsequent treatment trial that is less intense than 5+2 regimen according to physician/patient preference on study. Treatment continues in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection and bone marrow assessments on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Collection; Other: Electronic Health Record Review; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Collection — Undergo bone marrow assessment
  Other Names: Collection, Bone Marrow
Other: Electronic Health Record Review — Ancillary studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial studies whether less fit adults with acute myeloid leukemia (AML) or myeloid neoplasms are willing to let a computer program decide (randomization) whether they receive lower- or higher-intensity chemotherapy. Historically, treatment decision-making for patients with AML or myeloid neoplasms has divided patients into two categories, with patients considered fit receiving intensive "curative" chemotherapy, and patients considered unfit, such as older patients with a higher risk of early death from therapy, receiving non-intensive "palliative" therapy or no therapy. With the introduction of new treatment agents, it has become difficult to determine the difference between intensive and non-intensive therapy, especially for patients considered unfit for whom treatment-related side effects remain a concern. Treatment intensity is best identified through randomized trials but often patients are unwilling to undergo randomization due to preset beliefs. However, with improved supportive care and the awareness that new treatment agents may have similar risks as intensive therapy, it may be possible that more patients are willing to be randomized. This may help identify the best treatment intensity for less fit adults with AML or myeloid neoplasms, which may improve outcomes.

DETAILED DESCRIPTION:
OUTLINE:

This pilot umbrella trial will explore the feasibility of randomizing patients to higher or lower intensity treatment regimens.

The exact treatment regimens given will be at the discretion of the treating physician and will be provided either as standard of care or following enrollment on a subsequent treatment trial.

Patients and physicians indicate willingness to randomize, those willing are randomized to 1 of 2 arms, those unwilling choose arm III or IV.

ARM I: Patients receive standard of care (SOC) or investigational higher-intensity therapy on a subsequent treatment trial that is at least as intense as seven days of cytarabine in combination with three days of anthracycline (7+3 regimen) at the discretion of the treating physician on study. Treatment continues in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive SOC or investigational lower-intensity therapy on a subsequent treatment trial that is less intense than five days of cytarabine in combination with two days of anthracycline (5+2 regimen) at the discretion of the treating physician on study. Treatment continues in the absence of disease progression or unacceptable toxicity.

ARM III: Patients receive SOC or investigational higher-intensity therapy on a subsequent treatment trial that is at least as intense as 7+3 regimen according to physician/patient preference on study. Treatment continues in the absence of disease progression or unacceptable toxicity.

ARM IV: Patients receive SOC or investigational lower-intensity therapy on a subsequent treatment trial that is less intense than 5+2 regimen according to physician/patient preference on study. Treatment continues in the absence of disease progression or unacceptable toxicity.

Additionally, all patients undergo blood sample collection and bone marrow assessments on study.

After completion of study treatment, patients are followed up periodically for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of high grade myeloid neoplasm (> 10% blasts in blood or marrow), other than acute promyelocytic leukemia (APL) according to the 2022 International Consensus Classification (ICC) classification. Patients with acute leukemias of ambiguous lineage are eligible
* The use of cytoreductive therapy before treatment is permitted. Patients with symptoms/signs of leukostasis, white blood cell (WBC) > 100,000/μL, or acute symptoms that in the opinion of the treating physician are likely related to their high-grade myeloid neoplasm may receive up to 2 doses of cytarabine (up to 500 mg/m^2 each) prior to study day 1
* Patients may have received treatment for antecedent low-grade myeloid neoplasm (< 10% myeloid blasts on blood or bone marrow)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 3 (for patients aged < 75 years) or ECOG performance status of 0 - 2 (for patients aged ≥ 75 years)
* The presence of one or more of the following criteria for 'unfitness'. (Patients without respiratory symptoms at rest are eligible and should only complete spirometry/diffusion capacity of the lung for carbon monoxide [DLCO] measurements as clinically indicated):

  * ECOG Performance Status of 2 or 3
  * Cardiac history of congestive heart failure (CHF) requiring treatment or ejection fraction ≤ 50% or chronic stable angina
  * Documented DLCO ≤ 65% or forced expiratory volume in 1 second (FEV1) ≤ 65%; or dyspnea at rest, or requiring supplemental oxygen
  * Creatinine clearance ≥ 30 mL/min to < 45 ml/min
  * Moderate hepatic impairment with total bilirubin > 1.5 to ≤ 3.0 × upper limit of normal (ULN)
  * Any other comorbidity that the physician judges to be incompatible with intensive chemotherapy
* Adequate cardiac function:

  * Patients aged ≤ 60 years without a history of cardiac disease or evidence of heart failure are eligible if they also exhibit the following:

    * Chest x-ray (CXR) without evidence of moderate or severe pulmonary edema or pleural effusion, and a normal cardio-mediastinal silhouette
    * Electrocardiogram (ECG) without evidence of atrial or ventricular chamber enlargement
    * Note that patients with either abnormal CXR or ECG should have a structural heart assessment (echocardiogram, multigated acquisition scan [MUGA] or similar) and are eligible if left ventricular ejection fraction (LVEF) > 40% and the abnormalities in the CXR/ECG do not preclude safe administration of intensive chemotherapy
  * Patients with a documented left ventricular ejection fraction (LVEF) ≥ 40%, assessed within 3 months prior to registration, e.g. by MUGA scan or echocardiography, or another appropriate diagnostic modality are eligible
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3x ULN, unless judged due to leukemic organ involvement
* Total bilirubin ≤ 3 x ULN unless judged due to leukemic organ involvement, Gilbert's syndrome, or hemolysis
* Women of childbearing potential and men must agree to use adequate contraception beginning at the signing of the consent until at least 4 weeks after the last dose of study drug
* HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Known hypersensitivity to cytarabine, anthracycline, hypomethylating agents, or venetoclax
* Cardiovascular disability status of New York Heart Association class ≥ 2. Class 2 is defined as cardiac disease in which patients are comfortable at rest but ordinary physical activity results in fatigue, palpitations, dyspnea, or anginal pain
* Subject exhibits evidence of other clinically significant uncontrolled systemic infection requiring therapy (viral, bacterial or fungal)
* Concomitant illness associated with a likely survival of < 1 year
* Active pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Willingness to randomize (Feasibility) | At baseline
  Patient willingness to randomize will be indicated on the survey instrument Patient Preference for Treatment Assignment Survey. Patients who select the box indicating "I am willing to let a coin flip (i.e. computer program) decide whether I receive lower- or higher-intensity chemotherapy" will be considered willing to randomize. Will consider randomization feasible (i.e. a subsequent, larger study would be designed as a randomized trial) if the true proportion of patients willing to be randomized is 60% or higher.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Appelbaum, MD, PhD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No